CLINICAL TRIAL: NCT07209098
Title: Broaden Accessibility of Breakthrough Treatment for Heart Failure: A Prospective, Propensity-Matched CED to Access the Impact of Cardiac Contractility Modulation Therapy (CCM)
Brief Title: Propensity-Matched Study of Cardiac Contractility Modulation Therapy in Heart Failure
Acronym: BRIGHTEN-HF
Status: Recruiting | Type: Observational
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: CA_CP_2558
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure and Reduced Ejection Fraction; NYHA Class III Heart Failure
Keywords: Heart failure; Reduced ejection fraction; Cardiac Contractility Modulation; CCM; NYHA III; Propensity Score Matching; All-Cause Mortality; Heart Failure Hospitalizations; CED
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Treatment Group: Treatment patients shall be those with a clinical indication for CCM implantation according to FDA approved labeling and who are implanted with the Optimizer System.
  Interventions: Device: Cardiac Contractility Modulation (CCM)
- Control Group: The control group shall be derived from propensity score matching of patients derived from the database with a clinical indication for CCM implantation who do not receive an implant.

INTERVENTIONS:
Device: Cardiac Contractility Modulation (CCM) — CCM is a therapy delivered via the Optimizer System, which is implanted in eligible heart failure patients. The device delivers non-excitatory electrical signals to the heart during the absolute refractory period, enhancing the strength of cardiac contractions without increasing myocardial oxygen consumption.
  Groups: Treatment Group

SUMMARY:
The purpose of this prospective, multi-center, propensity-matched coverage with evidence development (CED) study is to assess the impact of cardiac contractility modulation (CCM) on mortality and heart failure hospitalizations in Medicare-eligible patients with heart failure who meet indications for CCM.

DETAILED DESCRIPTION:
Data for both the CCM treatment arm and a propensity-matched control group come from a large, de-identified, aggregated electronic health record (EHR) database containing patient information from multiple U.S. healthcare systems. The database includes demographics, clinical notes, imaging, laboratory results, medications, social determinants of health, and other relevant healthcare information, with up to 8 years of historical clinical data updated regularly.

ELIGIBILITY:
Inclusion Criteria

1. Continuous representation in the database in the year prior to index.
2. Age 18 or older will be enrolled in either the treatment or control arm of the study.
3. NYHA III heart failure,
4. Not receiving CRT
5. EF 25 - 45%, inclusive.
6. Remain symptomatic despite at least 3 months of optimized guideline-directed medical therapy (GDMT) as determined by the heart team prior to CCM implantation.

Exclusion Criteria

1. Subject has had a prior heart transplant
2. Subject with mechanical tricuspid valve.
3. Subject has a left ventricular assist device (LVAD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients with heart failure who are identified from a large, de-identified, multi-system electronic health record (EHR) database representing diverse healthcare settings across the United States. The database includes patients receiving care in hospitals, outpatient clinics, and other sites where cardiac contractility modulation (CCM) therapy is delivered. The population reflects typical sites of CCM implantation in Medicare-eligible adults across multiple states and integrated delivery networks (IDNs).
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Time to first heart failure hospitalization or all-cause death | Up to 2 years post-index date for each patient; follow-up will continue until 2 years after the last patient is enrolled to allow at least 2 years of observation for all participants.
  Time from index date to the first occurrence of either heart failure-related hospitalization or death in patients with a clinical indication for cardiac contractility modulation (CCM) therapy. Outcomes will be compared between patients implanted with the Optimizer System (treatment arm) and a propensity score-matched control group of patients who are eligible for CCM but did not receive the device. Data will be collected from a large, de-identified, multi-system electronic health record database representing diverse sites of care across the United States.

OTHER OUTCOMES:
Time to recurrent heart failure hospitalization | Up to 2 years post-index date for each patient; follow-up continues until 2 years after the last patient is enrolled to allow at least 2 years of observation.
  Time from index date (CCM implantation for treatment patients) to each heart failure-related hospitalization, including first and subsequent hospitalizations, in patients receiving CCM therapy compared with a matched control group of patients eligible for CCM but not treated. This outcome is exploratory and hypothesis-generating.
Time to all-cause mortality | Up to 2 years post-index date for each patient; follow-up continues until 2 years after the last patient is enrolled to allow at least 2 years of observation.
  Time from index date (CCM implantation for treatment patients) to death from any cause, in patients receiving CCM therapy compared with a matched control group of patients eligible for CCM but not treated. This outcome is exploratory and hypothesis-generating.

CONTACTS AND LOCATIONS:
Locations (1):
- Impulse Dynamics, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided